CLINICAL TRIAL: NCT04731363
Title: Consumption of Oral Artificial Sweeteners on Platelet Aggregation and Polyol Excretion
Acronym: COSETTE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff, Cellular and Molecular Medicine & Cardiovascular Medicine, Section of Heart Failure, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-005
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: xylitol; erythritol
MeSH Terms: interventions — Xylitol; Erythritol; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Xylitol, 30g (Experimental): oral xylitol, a potent artificial sweetener
  Interventions: Dietary Supplement: xylitol, 30g
- Erythritol, 30g (Experimental): oral erythritol, a potent artificial sweetener
  Interventions: Dietary Supplement: erythritol, 30g
- Xylitol, 5g (Experimental): oral xylitol, a potent artificial sweetener
  Interventions: Dietary Supplement: xylitol, 5g
- Glucose, 30g (Active Comparator): oral glucose, delivered as dextrose
  Interventions: Dietary Supplement: glucose, 30g

INTERVENTIONS:
Dietary Supplement: xylitol, 30g — Intervention is a drink consisting of 300mL of water containing 30g of xylitol as a single oral dose.
  Arms: Xylitol, 30g
Dietary Supplement: erythritol, 30g — Intervention is a drink consisting of 300mL of water containing 30g of erythritol as a single oral dose.
  Arms: Erythritol, 30g
Dietary Supplement: xylitol, 5g — Intervention is a drink consisting of 300mL of water containing 5g of xylitol as a single oral dose.
  Arms: Xylitol, 5g
Dietary Supplement: glucose, 30g — Intervention is a drink consisting of 300mL of water containing 30g of glucose (dextrose) as a single oral dose.
  Other Names: dextrose, 30g
  Arms: Glucose, 30g

SUMMARY:
The principal goal for the study is to examine whether ingestion of a beverage containing artificial sweeteners alters in vitro platelet aggregation.

Because of the increasing number of cardiometabolic diseases, such as diabetes mellitus, in the population, the use of artificial sweeteners to replace free sugars has been gaining popularity. Two popular artificial sweeteners are erythritol and xylitol. Erythritol and xylitol are both naturally occurring polyols found in fruits and vegetables. They are potent artificial sweeteners with a higher sweetening intensity and lower calorie content than table sugar.

Previous research has shown that the higher levels of sugar alcohols, like those used as artificial sweeteners, in the blood are related to a higher risk of cardiovascular complications, like heart attacks and strokes, and death. This may be because higher levels of sugar alcohols in one's blood may increase the activity of platelets, which would then increase the risk of heart attack and stroke. The investigators therefore want to find if consuming a single beverage that contains an artificial sweetener can raise the levels of sugar alcohols in the blood and if it can alter platelet function or aggregation.

DETAILED DESCRIPTION:
The purpose of this study is to examine if drinking a single beverage that contains an artificial sweetener can perceptibly alter the activity of platelets in the body. Platelets are a component of blood that are primarily responsible for helping to stop bleeding and repair damaged blood vessels by grouping together, a process known as aggregation, to form clots.

Artificial sweeteners are popular because they have a lower calorie content than table sugar while still making food and beverages sweet. Their use as a sugar substitute is especially attractive for people with heart disease or diabetes, or for people who are trying to lose weight.

Two popular artificial sweeteners are erythritol and xylitol. Erythritol and xylitol are both naturally occurring polyols, also called sugar alcohols, found in fruits and vegetables. They are potent artificial sweeteners with a higher sweetening intensity and lower calorie content than table sugar.This makes them attractive for the use as sugar substitutes or alternatives, particularly for patients with type 2 diabetes.

Up to now, there is no prospective data available about polyols with respect to their impact on event outcomes in cardiovascular patients, despite their extensive use in the food industry. Moreover, little is known about plasma levels and metabolic changes following food intake of artificial sweeteners, in particular polyols.

The investigators have previously measured fasting levels of various polyols in a large clinical cohort of cardiovascular patients and found that some candidate polyols are related to a higher risk of cardiovascular complications and death. In vitro data using human platelets revealed that the polyols xylitol and erythritol at the levels observed in fasting patients induce platelet aggregation potential. The investigator's data shows that erythritol and xylitol impact platelet function and may, therefore, contribute to cardiovascular mortality.

In preliminary studies the investigators found that when ingesting either erythritol or xylitol, the levels of these sweeteners in the plasma rise within the first hour after consumption. With this study the investigators wish to examine whether the postprandial levels are capable of altering platelet function in vitro. The investigators hypothesize that postprandial polyol concentrations following ingestion increase platelet aggregation in the blood.

ELIGIBILITY:
Cohort 1 Inclusion Criteria:

* Age 18 years or above.
* Willing and able to sign the consent form.

Cohort 1 Exclusion Criteria:

* Use of anti-platelet medications within 14 days of study enrollment.
* Active infection or received antibiotics within 1 month of study enrollment.
* Use of over-the-counter probiotic within 1 month of study enrollment.
* Diabetes mellitus
* Ulcerative colitis, Crohn's disease, or other chronic gastrointestinal disorder.
* Past history of bariatric procedures or surgeries (e.g. gastric banding or bypass).
* Pregnancy.
* Significant chronic illness.

Cohort 2 Inclusion Criteria:

* Men and women age 18 years or above.
* Able to provide informed consent and comply with study protocol.
* Diabetes Mellitus Type II

Cohort 2 Exclusion Criteria:

* Use of anti-platelet medications within 14 days of study enrollment.
* Active infection or received antibiotics within 1 month of study enrollment.
* Use of over-the-counter probiotic within 1 month of study enrollment.
* Ulcerative colitis, Crohn's disease, or other chronic gastrointestinal disorder.
* Past history of bariatric procedures or surgeries (e.g. gastric banding or bypass).
* Pregnancy.
* Any condition that, in the judgment of the Investigator, would place a subject at undue risk by being enrolled in the trial or cause inability to comply with the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makinen KK. Gastrointestinal Disturbances Associated with the Consumption of Sugar Alcohols with Special Consideration of Xylitol: Scientific Review and Instructions for Dentists and Other Health-Care Professionals. Int J Dent. 2016;2016:5967907. doi: 10.1155/2016/5967907. Epub 2016 Oct 20. PMID 27840639
- [Background] Oku T, Okazaki M. Laxative threshold of sugar alcohol erythritol in human subjects. Nutrition Research. 1996;16(4):577-89.
- [Result] Witkowski M, Nemet I, Alamri H, Wilcox J, Gupta N, Nimer N, Haghikia A, Li XS, Wu Y, Saha PP, Demuth I, Konig M, Steinhagen-Thiessen E, Cajka T, Fiehn O, Landmesser U, Tang WHW, Hazen SL. The artificial sweetener erythritol and cardiovascular event risk. Nat Med. 2023 Mar;29(3):710-718. doi: 10.1038/s41591-023-02223-9. Epub 2023 Feb 27. PMID 36849732
- [Result] Witkowski M, Nemet I, Li XS, Wilcox J, Ferrell M, Alamri H, Gupta N, Wang Z, Tang WHW, Hazen SL. Xylitol is prothrombotic and associated with cardiovascular risk. Eur Heart J. 2024 Jul 12;45(27):2439-2452. doi: 10.1093/eurheartj/ehae244. PMID 38842092
- [Result] Witkowski M, Wilcox J, Province V, Wang Z, Nemet I, Tang WHW, Hazen SL. Ingestion of the Non-Nutritive Sweetener Erythritol, but Not Glucose, Enhances Platelet Reactivity and Thrombosis Potential in Healthy Volunteers-Brief Report. Arterioscler Thromb Vasc Biol. 2024 Sep;44(9):2136-2141. doi: 10.1161/ATVBAHA.124.321019. Epub 2024 Aug 8. PMID 39114916

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Started | 10 | 25 | 5 | 10
Completed | 10 | 23 | 5 | 10
Not Completed | 0 | 2 | 0 | 0
Not completed — Could not obtain samples | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g | Total
Number analyzed (Participants) | 10 | 23 | 5 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.1) | 35.8 (14.0) | 31.2 (10.1) | 30.1 (11.5) | 34.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 3 | 6 | 26
  Male | 5 | 11 | 2 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 22 | 5 | 9 | 46
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 2 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2 | 4
  White | 8 | 16 | 3 | 6 | 33
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 23 | 5 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: Platelet Aggregation After Polyol Ingestion
Description: Measuring platelet function 30 minutes after polyol ingestion, using established in vitro platelet assays. Platelet aggregation responses, based on changes in light transmission after adding different concentrations of the agonists ADP and TRAP6 are reported. A higher percentage of light transmission indicates an increased aggregation response, with maximum amplitude (100%) indicating total aggregation.
Time Frame: 30 minutes
Population: Only 10 of the 23 subjects consuming 30g of erythritol had aggregometry measurements performed. These were the last 10 subjects enrolled in this arm. The earlier subjects were only used to assess levels of erythritol following ingestion (pharmacokinetics studies) without looking at platelet function. The pharmacokinetics studies informed the subsequent aggregometry experiments in the final 10 subjects.
Measure: Median (Inter-Quartile Range); unit: % of maximum amplitude
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 10 | 5 | 10
% of maximum amplitude
  ADP (1 uM) | 20.00 [16.00 to 25.00] | 18.50 [14.25 to 23.00] | 20.00 [16.25 to 23.00] | 12.00 [10.00 to 13.75]
  ADP (2 uM) | 33.00 [30.00 to 40.00] | 34.00 [29.00 to 39.50] | 29.00 [23.00 to 33.00] | 22.00 [20.00 to 24.00]
  ADP (3 uM) | 43.50 [41.00 to 61.00] | 42.50 [37.00 to 52.00] | 44.00 [39.00 to 48.00] | 31.00 [27.00 to 33.00]
  ADP (4 uM) | 57.00 [53.00 to 70.00] | 66.50 [55.00 to 70.75] | 72.50 [63.75 to 77.25] | 49.00 [45.50 to 56.50]
  TRAP6 (2.5uM) | 13.00 [9.50 to 24.00] | 15.00 [8.00 to 21.25] | 9.00 [5.00 to 17.00] | 1.00 [0.00 to 3.00]
  TRAP6 (5.0uM) | 32.00 [19.00 to 49.00] | 26.00 [17.50 to 38.00] | 16.50 [10.75 to 26.00] | 8.00 [5.50 to 12.00]
  TRAP6 (7.5 uM) | 50.00 [37.50 to 72.50] | 45.00 [34.00 to 53.50] | 37.00 [29.00 to 60.00] | 20.00 [18.00 to 23.00]
  TRAP6 (10.0uM) | 68.00 [59.50 to 73.50] | 69.00 [64.00 to 75.00] | 78.00 [67.00 to 86.00] | 61.00 [51.50 to 65.50]

2. Primary Outcome: Change From Baseline in Platelet Aggregation at 30 Minutes Post Polyol Ingestion
Description: Measuring changes in platelet function before versus after xylitol or erythritol ingestion, using established in vitro platelet assays. Platelet aggregation responses, based on changes in light transmission after adding different concentrations of the agonists ADP and TRAP6 are reported. A higher percentage of light transmission indicates an increased aggregation response, with maximum amplitude (100%) indicating total aggregation.
Time Frame: Baseline and 30 minutes post ingestion of polyol intervention
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: % of maximum amplitude
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 10 | 5 | 10
% of maximum amplitude
  1uM ADP at Baseline | 11.00 [9.00 to 13.00] | 11.00 [9.00 to 13.00] | 11.00 [8.00 to 13.00] | 11.50 [9.00 to 13.00]
  1uM ADP at 30 minutes post polyol ingestion | 20.00 [16.00 to 25.00] | 18.50 [14.25 to 23.00] | 20.00 [16.25 to 23.00] | 12.00 [10.00 to 13.75]
  2 uM ADP at Baseline | 21.00 [19.00 to 23.00] | 22.00 [18.00 to 25.00] | 19.00 [16.00 to 24.00] | 21.00 [18.00 to 23.00]
  2 uM ADP at 30 minutes post polyol ingestion | 33.00 [30.00 to 40.00] | 34.00 [29.00 to 39.50] | 29.00 [23.00 to 33.00] | 22.00 [20.00 to 24.00]
  3uM ADP at Baseline | 30.00 [28.00 to 31.75] | 30.00 [28.00 to 34.00] | 31.00 [28.00 to 33.00] | 30.00 [28.00 to 32.00]
  3uM ADP at 30 minutes post polyol ingestion | 43.50 [41.00 to 61.00] | 42.50 [37.00 to 52.00] | 44.00 [39.00 to 48.00] | 31.00 [27.00 to 33.00]
  4uM ADP at Baseline | 45.00 [38.00 to 50.00] | 50.50 [46.00 to 57.75] | 52.00 [47.00 to 54.50] | 50.00 [46.00 to 53.50]
  4uM ADP at 30 minutes post polyol ingestion | 57.00 [53.00 to 70.00] | 66.50 [55.00 to 70.75] | 72.50 [63.75 to 77.25] | 49.00 [45.50 to 56.50]
  2.5 uM TRAP6 at Baseline | 2.50 [1.00 to 4.00] | 2.50 [1.00 to 3.25] | 2.00 [0.00 to 4.00] | 1.00 [0.00 to 3.00]
  2.5 uM TRAP6 at 30 minutes post polyol ingestion | 13.00 [9.50 to 24.00] | 15.00 [8.00 to 21.25] | 9.00 [5.00 to 17.00] | 1.00 [0.00 to 3.00]
  5.0 uM TRAP6 at Baseline | 9.00 [8.00 to 12.00] | 9.00 [7.00 to 12.00] | 9.00 [7.00 to 10.25] | 9.00 [8.00 to 11.00]
  5.0 uM TRAP6 at 30 minutes post polyol ingestion | 32.00 [19.00 to 49.00] | 26.00 [17.50 to 38.00] | 16.50 [10.75 to 26.00] | 8.00 [5.50 to 12.00]
  7.5 uM TRAP6 at Baseline | 20.00 [17.00 to 23.50] | 20.00 [17.00 to 23.00] | 21.00 [18.00 to 25.00] | 19.00 [17.00 to 22.00]
  7.5 uM TRAP6 at 30 minutes post polyol ingestion | 50.00 [37.50 to 72.50] | 45.00 [34.00 to 53.50] | 37.00 [29.00 to 60.00] | 20.00 [18.00 to 23.00]
  10.0 uM TRAP6 at Baseline | 45.50 [40.00 to 50.00] | 48.00 [45.00 to 54.00] | 60.00 [46.00 to 64.00] | 61.50 [58.50 to 65.00]
  10.0 uM TRAP6 at 30 minutes post polyol ingestion | 68.00 [59.50 to 73.50] | 69.00 [64.00 to 75.00] | 78.00 [67.00 to 86.00] | 61.00 [51.50 to 65.50]

3. Primary Outcome: Plasma Polyol Levels After Polyol Ingestion
Description: Measuring plasma levels (uM) of polyols (xylitol or erythritol) 30 minutes after xylitol or erythritol ingestion, using established techniques by mass spectrometry. Xylitol was measured, and is reported below, in the two xylitol intervention arms and erythritol was measured, and is reported below, in the erythritol and glucose intervention arms.
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 23 | 5 | 10
uM | 312.4 [133.9 to 628.5] | 6174.9 [5546.5 to 7034.3] | 0.97 [0.95 to 1.43] | 2.9 [2.7 to 3.8]

4. Primary Outcome: Change From Baseline in Plasma Polyol Levels at 30 Minutes Post Polyol Ingestion
Description: Measuring changes in levels of plasma polyols before versus after xylitol or erythritol ingestion, using established techniques by mass spectrometry. Xylitol concentrations are reported in the two xylitol intervention arms. Erythritol concentrations are reported in the erythritol and glucose intervention arms.
Time Frame: Baseline and 30 minutes post ingestion of polyol intervention
Measure: Median (Inter-Quartile Range); unit: umol/L (uM)
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 23 | 5 | 10
umol/L (uM)
  Baseline | 0.30 [0.27 to 0.34] | 3.8 [3.5 to 4.1] | 0.26 [0.23 to 0.38] | 3.0 [2.6 to 4.0]
  30 minutes post-ingestion of polyol | 312.4 [133.9 to 628.5] | 6174.9 [5546.5 to 7034.3] | 0.97 [0.95 to 1.43] | 2.9 [2.7 to 3.8]

5. Primary Outcome: Urinary Polyol Levels After Polyol Ingestion
Description: Measuring the urinary levels of polyols (xylitol or erythritol) 30 minutes after xylitol or erythritol ingestion, using established techniques by mass spectrometry. Xylitol was measured, and is reported below, in the two xylitol intervention arms and erythritol was measured, and is reported below, in the erythritol and glucose intervention arms.
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 23 | 5 | 10
uM | 5242.00 [1500.06 to 16662.00] | 86832.00 [64506.00 to 162204.00] | 29.20 [9.88 to 75.84] | 225.56 [92.32 to 471.78]

6. Primary Outcome: Change From Baseline in Urinary Polyol Levels at 30 Minutes Post Polyol Ingestion
Description: Measuring changes in levels of urinary polyols before versus after xylitol or erythritol ingestion, using established techniques by mass spectrometry. Xylitol was measured, and is reported below, in the two xylitol intervention arms and erythritol was measured, and is reported below, in the erythritol and glucose intervention arms.
Time Frame: Baseline and 30 minutes post ingestion of polyol intervention
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 10 | 23 | 5 | 10
uM
  Baseline | 42.24 [27.32 to 51.90] | 372.56 [220.70 to 566.76] | 18.92 [5.36 to 59.72] | 393.84 [260.49 to 629.45]
  30-minutes Post Polyol Ingestion | 5242.00 [1500.06 to 16662.00] | 86832.00 [64506.00 to 162204.00] | 29.20 [9.88 to 75.84] | 225.56 [92.32 to 471.78]

7. Secondary Outcome: Change From Baseline in Plasma Lipid Profile at 1 Day Post Polyol Ingestion
Description: Measuring changes in lipid levels as markers of changes in metabolism before versus after xylitol or erythritol ingestion.
Time Frame: Baseline and 1 day post ingestion of polyol intervention
Population: Not all subjects had blood drawn at 1 day post-sweetener ingestion. Blood samples at 1 day post ingestion were only obtained from 13 subjects who consumed 30g erythritol and 4 subjects who consumed 30g of xylitol. No subjects taking glucose or 5mg of xylitol had blood drawn at 1 day post-ingestion.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
Number analyzed (Participants) | 4 | 13 | 0 | 0
mg/dL
  Total Cholesterol at Baseline | 218.5 [207.8 to 226.0] | 168.0 [143.0 to 192.0] |  |
  Total Cholesterol at 1 day Post Polyol Ingestion | 203.5 [200.5 to 217.0] | 168.0 [145.0 to 199.0] |  |
  HDL at Baseline | 50.6 [46.7 to 57.8] | 51.6 [49.2 to 64.9] |  |
  HDL at 1 day Post Polyol Ingestion | 48.4 [46.0 to 56.7] | 52.4 [47.7 to 61.9] |  |
  Triglycerides at Baseline | 108.5 [93.0 to 133.5] | 80.0 [59.0 to 104.0] |  |
  Triglycerides at 1 day Post Polyol Ingestion | 106.0 [81.8 to 132.3] | 86.0 [63.0 to 103.0] |  |
  Calculated LDL at Baseline | 112.2 [55.0 to 170.2] | 91.0 [75.0 to 116.0] |  |
  Calculated LDL at 1 day Post Polyol Ingestion | 134.0 [123.5 to 148.8] | 97.0 [76.0 to 122.0] |  |

ADVERSE EVENTS:
Time Frame: Adverse events data was collected duration of enrollment period (1-12 days for each subject depending on arm assignment).
Arm/Group | Xylitol, 30g | Erythritol, 30g | Xylitol, 5g | Glucose, 30g
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/25 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/25 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/25 | 0/5 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04731363/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT04731363/SAP_001.pdf